CLINICAL TRIAL: NCT03791177
Title: The Effects of Listening to Music on Anxiety, Pain and Satisfaction During Urodynamic Study : A Randomized Controlled Trial
Brief Title: Urodynamics and Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Gül, Assistant Professor, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AksarayUTRH2
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Incontinence, Urinary
Keywords: Music
MeSH Terms: conditions — Urinary Incontinence | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The trial was blinded for data manager ( a nurse collecting the control and study group data) and statistician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): A total of 70 patients were included in the study. Using simple randomization method, the patients were acknowledged about the aim of the study and the cards with letters C (control) and S (study) were placed in closed envelopes and the patients were asked to draw a random envelope. After the draw, two groups were formed according to the letter as group I consisted of patients with C letter and group II consisted of patients with S letter.
  Interventions: Other: Music Therapy
- Control Group (Sham Comparator): A total of 70 patients were included in the study. Using simple randomization method, the patients were acknowledged about the aim of the study and the cards with letters C (control) and S (study) were placed in closed envelopes and the patients were asked to draw a random envelope. After the draw, two groups were formed according to the letter as group I consisted of patients with C letter and group II consisted of patients with S letter.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — Patients in the study group were exposed to flute music therapy (Sufi musical recital - Huseyni mode) at low tempo (60-80 rhythm / min) with weak beats and calm rhythms during the UDS.
  This audition involves both vocal and instrumental music performed by a reed flute called 'Ney'. A competent lecturer who was specialized in music suggested all the musical compositions during the therapy

SUMMARY:
Today music acts as an analgesic and anxiolytic in a safe, cheap and simple way. Several trials have confirmed its potential administration and benefits in urology practice. We aimed to assess the influence of music therapy on perceived anxiety and pain during outpatient urodynamic study (UDS) using the Visual Analog Scale (VAS) and the State-Trait Anxiety Inventory (STAI) in a prospective, randomized fashion

DETAILED DESCRIPTION:
Urodynamic study (UDS) is often used to help urologists to evaluate the functions of bladder and urethra in outpatient clinic.1 Although a UDS is a reliable tool for accurate diagnosis, the process itself can be accompanied by discomfort and pain as it includes the positioning the catheters urethral and rectally, and the bladder filling. Reports of having such invasive outpatient process whilst awake may demonstrate pain and disquiet that result in incomplete examinations and patient noncompliance2,3.

Various pharmacologic options including lidocaine gel and catheter tip lubrication for urethral catheterization were used to relieve pain and anxiety during UDS. Besides, there are some non-pharmalogical methods such as patient education, heating pad, music, distraction and relaxation4-6.

Music has been considered complementary treatment modality as cheap, safe and effective. In various urological procedures including cystoscopy, transrectal prostate biopsy and extracorporeal shock wave lithotripsy (ESWL) music has been proven helpful on pain and anxiety levels 7-10. However, current literature presents limited and controversial data evaluating the influence of music on pain and anxiety perspective of the patient during UDS. We, therefore, aimed to assess the effect of music on patient satisfaction in a analgesic and anxiolytic way during UDS.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Exclusion criteria included paraplegia, hearing impairment, taking any analgesic or anxiolytic drug to suppress the symptoms of anxiety until 24 hours prior to UDS, inability to understand or fulfill commands during UDS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Pain Scale: VAS | 10 minutes after UDS
Anxiety Scale: STAI | 10 minutes after UDS

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University Training and Research Hospital, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No